CLINICAL TRIAL: NCT05292274
Title: NIH RECOVER: A Multi-site Pathology Study of Post-Acute Sequelae of SARS-CoV-2 Infection
Brief Title: NIH RECOVER Tissue Pathology: Understanding the Long-Term Impact of COVID-19
Status: Recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: RECOVER-Path
Record Dates: First submitted 2022-03-22; First posted 2022-03-23 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: COVID-19; SARS CoV 2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — blood, body fluids, snap frozen and formalin-fixed tissue samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Post-Acute Sequelae of SARS-CoV-2 (PASC) Autopsy Study is a cross-sectional study designed to define and characterize the epidemiology, natural history, clinical spectrum, and underlying mechanisms of post-acute effects of SARS-CoV-2 infection in a diverse population representative of the general COVID-19 population in the US. The autopsy study will characterize the pathology of PASC in (i) non-hospitalized patients who die 30 days or later from symptom onset of COVID-19, and (ii) hospitalized patients who die 30 days or later after discharge from a hospitalization for COVID-19. The study will include decedents who had previously fully recovered from SARS-CoV-2 infection (i.e., >30 days from onset in non-hospitalized, or >30 days from discharge in hospitalized patients), and decedents who meet clinical criteria of PASC as defined by the recent World Health Organization publication (see Section 5.4 below). The autopsy study will also explore the pathology of acute SARS-CoV-2 infection in a smaller subset of patients who died 15-30 days from symptom onset. This protocol defines the common set of clinical data elements, autopsy procedures for tissue collection, core measures, pathology protocols, shared pathology tissues, data elements, and methodology. Each investigator site is expected to perform autopsies on the decedents to address the pathophysiology of the potential long-term effects of SARS-CoV-2 infection on human health. The Consortium analysis plan aims to address research questions by incorporating: 1) tissue obtained from autopsies performed at each Phase II participant's site; and 2) tissue available from other pathology investigators/autopsy sites within the Consortium.

ELIGIBILITY:
Inclusion Criteria:

Patients with suspected SARS-CoV-2 infection

1. Patients who meet the clinical and epidemiological criteria listed below:

   Clinical criteria: Acute onset of fever and cough or acute onset of ANY THREE OR MORE of the following signs or symptoms: fever, cough, general weakness/fatigue, headache, myalgia, sore throat, coryza, dyspnea, anorexia/nausea/vomiting, diarrhea, altered mental status.

   Epidemiological criteria:
   1. Having resided or worked in an area with a high risk of transmission of virus: closed residential, school, or camp settings any time within the 14 days before symptom onset; or
   2. Having resided or traveled to an area with community transmission any time within the 14 days before symptom onset; or
   3. Any known household contact or any member of the household working in any health care setting, including within health facilities or within the community, any time within the 14 days before symptom onset.
2. An asymptomatic person not meeting epidemiologic criteria with a positive SARS-CoV-2 Antigen-RDT.

Patients with probable SARS-CoV-2 infection

1. A patient who meets clinical criteria above AND is a contact of a probable or confirmed case or linked to a COVID-19 cluster; or
2. A suspected case with chest imaging showing findings suggestive of COVID-19 disease; or
3. A person with recent onset of anosmia (loss of smell) or ageusia (loss of taste) in the absence of any other identified cause; or
4. Death, not otherwise explained, in an adult with respiratory distress preceding death AND who was a contact of a probable or confirmed case or linked to a COVID-19 cluster.

Patients with confirmed SARS-CoV-2 infection

1. A person with a positive Nucleic Acid Amplification Test (NAAT); or
2. A person with a positive SARS-CoV-2 Antigen-RDT AND meeting either the probable case definition or suspected criteria a) or b); or
3. An asymptomatic person with a positive SARS-CoV-2 Antigen-RDT who was a contact of a probable or confirmed case.

General Eligibility Notes:

1. Decedents with or without history of MIS-A or MIS-C are eligible;
2. Decedents with or without history of SARS-CoV-2 vaccination are eligible;
3. Decedents with recurrent SARS-CoV-2 infections and those with post-vaccination (breakthrough) infections are eligible;
4. Decedents are eligible without exclusion related to sex, race/ethnicity, geography, nationality, severity of disease, or underlying health conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Decedents over the age of 18 years at the time of death will be eligible for inclusion. Infected individuals will have suspected, probable, or confirmed SARS-CoV-2 infection as defined by WHO criteria, within 24 months of enrollment.
  Next of kin will provide consent in accordance with local legal requirements to participate in autopsy and biological sample collection as specified in the protocol procedures.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2022-03-08 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Number of decedents with presence of inflammation | Month 24
  In decedents with acute SARS-CoV-2 infection (dying 15-30 days after infection), and in decedents with prior SARS-CoV-2 infection (who die more than 30 days after initial onset, in-hospital and out-of-hospital) with and without PASC.
Number of decedents with presence of fibrosis | Month 24
  In decedents with acute SARS-CoV-2 infection (dying 15-30 days after infection), and in decedents with prior SARS-CoV-2 infection (who die more than 30 days after initial onset, in-hospital and out-of-hospital) with and without PASC.
Number of decedents with presence of thrombosis | Month 24
  n decedents with acute SARS-CoV-2 infection (dying 15-30 days after infection), and in decedents with prior SARS-CoV-2 infection (who die more than 30 days after initial onset, in-hospital and out-of-hospital) with and without PASC.
Number of decedents with presence of necrosis | Month 24
  In decedents with acute SARS-CoV-2 infection (dying 15-30 days after infection), and in decedents with prior SARS-CoV-2 infection (who die more than 30 days after initial onset, in-hospital and out-of-hospital) with and without PASC.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Katz, MD, Principal Investigator — NYU Langone Health; Leora Horwitz, MD, Principal Investigator — NYU Langone Health; Andrea Troxel, ScD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Beginning 9 months and with no end date. Data products from this study will be made available to researchers and analysts through the PASC Consortium Data Resource Core.
Access Criteria: The investigator who proposed to use the data will have access upon reasonable request. Requests should be directed to RECOVER_CSC@NYULangone.org. To gain access, data requestors will need to sign a data access agreement.